CLINICAL TRIAL: NCT03280433
Title: Association of the Volume and Proteome of Epicardial Adipose Tissue With Coronary Artery Disease, Left Atrial Remodelling and Atrial Fibrillation in Severe Aortic Stenosis Patients
Brief Title: Influence of EPICardial Adipose Tissue in HEART Diseases: EPICHEART Study
Acronym: EPICHEART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government)
Collaborators: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Jennifer Mancio, Principal Investigator, Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E.
Other Study IDs: SFRH/BD/104369/2014
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease; Coronary Arteriosclerosis; Atrial Fibrillation; Left Atrial Abnormality; Severe Aortic Stenosis
Keywords: Epicardial adipose tissue; Coronary artery disease; Atrial fibrillation; Severe aortic stenosis; Proteome; Mass spectrometry; Computed tomography
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation; Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fat samples (Epicardial fat, mediastinal fat, and subcutaneous fat), blood samples, pericardial fluid samples, right atrial appendage sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Aortic valve replacement

SUMMARY:
This translational study was designed to explore the association of the quantity and quality of epicardial adipose tissue (EAT) with coronary artery disease (CAD), left atrial remodeling and postoperative atrial fibrillation in a high cardiovascular disease-risk population. The investigators expect to identify new biochemical factors and biomarkers in the crosstalk between the epicardial adipocytes, coronary plaques and atrial cardiomyocytes that are involved in the pathogenesis of atherosclerosis and atrial fibrillation, respectively.

DETAILED DESCRIPTION:
Background: EAT has emerged as a new independent, and, potentially, modifiable cardiovascular risk factor for CAD. EAT volume assessed by computed tomography (CT) was independently associated with the presence of coronary stenosis, coronary calcification and myocardial ischemia in cross-sectional studies, and, prospectively, with major adverse cardiovascular events. Most of these clinical studies were, however, derived from community-based patients with low-to intermediate-risk profile and the role of EAT in high-risk patients is currently unclear. Accumulation of EAT has been also associated with left atrial (LA) dilation, presence, chronicity, and recurrence of atrial fibrillation (AF). Although there is evidence suggesting that EAT may be a major determinant of the LA vulnerable substrate of AF, the mechanisms in the causal pathway between the EAT and LA remodeling are not completely elucidated.

Aims: The main aims are to investigate if the volume of the EAT on CT and EAT proteome assessed by SWATH-mass spectrometry are associated with extent, distribution and complexity of coronary stenosis and coronary artery calcification, left atrial strain and incidence of postoperative atrial fibrillation in patients with symptomatic severe aortic stenosis.

Methods: This a prospective study enrolling symptomatic severe aortic stenosis patients referred to aortic valve replacement. The protocol includes preoperative detailed clinical and nutritional evaluations, echocardiography, CT, cardiac magnetic resonance imaging and invasive coronary angiography. During cardiac surgery, biopsies from the EAT, mediastinal and subcutaneous thoracic adipose tissues will be performed to undergo analysis of proteome using SWAT-mass spectrometry. Samples from the pericardial fluid, circulating and coronary sinus blood samples will be collected as well in order to find local and peripheral adipose tissue-derived biomarkers of the disease.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic severe aortic stenosis patients (defined as aortic valve area of < 1 cm2 or 0.6 cm2/m2 by transthoracic echocardiography) referred to aortic valve replacement.

Exclusion Criteria:

* diagnosis of acute coronary syndrome in the last 3 months.
* prior history of persistent or permanent atrial or flutter fibrillation.
* coexisting moderate to severe aortic valve regurgitation or moderate to severe mitral valve disease, bicuspid aortic valve.
* left ventricular dilatation [end-diastolic volume index >75 mL/m²].
* left ventricular ejection fraction <55%.
* chronic renal failure stage 3 to 5 defined as glomerular filtration rate GFR estimated by Cockcroft-Gault formula adjusted for body surface area < 30 mL/min/1.73m².
* moderate to severe chronic obstructive pulmonary disease defined as forced expiratory volume in one second <50% according to the 2011 Global Initiative for Chronic Obstructive Pulmonary Disease guidelines.
* active malignancy (i.e. With no evidence of recurrence and no longer receiving active treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic severe aortic stenosis referred to aortic valve replacement.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2018-11-25 (Estimated)

PRIMARY OUTCOMES:
New onset atrial fibrillation | Intra-hospital (i.e. from surgery until hospital discharge which means 7 days on average)
  Incidence of atrial fibrillation after aortic valve replacement
Left atrial remodelling by transthoracic echocardiography and magnetic resonance imaging | 6-month following aortic valve replacement
  Change in left atrial strain and volumes
Frailty syndrome according to Fried et al. scale | 6-month following aortic valve replacement
  Change in frailty syndrome classification
Coronary artery disease according to the presence of coronary stenosis and/or calcification | Baseline
  Prevalent coronary artery stenosis and coronary calcification

SECONDARY OUTCOMES:
Left ventricular hypertrophy by transthoracic echocardiography and magnetic resonance imaging | 6-month following aortic valve replacement
  Regression of left ventricular mass after aortic valve replacement
Right ventricular structure and function by transthoracic echocardiography and magnetic resonance imaging | 6-month following aortic valve replacement
  Changes in right ventricular structure and function after aortic valve replacement

OTHER OUTCOMES:
Mortality | 3- to 5-year after aortic valve replacement
  Incidence of all-cause death after aortic valve replacement

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Porto District
  - Faculty of Medicine of Porto, Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baeza R, Nunes F, Santos C, Mancio J, Fontes-Carvalho R, Renna F, Pedrosa J. Validation of a deep learning approach for epicardial adipose tissue segmentation in computed tomography. Int J Cardiovasc Imaging. 2025 Nov 13. doi: 10.1007/s10554-025-03528-1. Online ahead of print. PMID 41233698